

# STATISTICAL ANALYSIS PLAN

Protocol Title: A Phase 2, Open-Label, Single-Arm Study of Single-

Dose Lead-In and Neoadjuvant Trilaciclib and Chemotherapy in Patients with Early-Stage Triple

**Negative Breast Cancer (TNBC)** 

**Protocol Version** 2.0

**Protocol Number:** G1T28-212

Compound: Trilaciclib for Injection, 300 mg/vial

Study Phase: Phase 2
Study Name: MOA

**Sponsor:** G1 Therapeutics, Inc.

**Legal Registered Address:** 700 Park Offices Dr. Suite 200

PO Box 110341

Research Triangle Park, NC 27709

**Regulatory Agency Identifier** 

**Numbers:** 

IND: 145091

V 2.0

**Statistical Analysis Plan** 

Version:

**Approval Date:** 18 Apr 2023

#### SAP SIGNATURE PAGE

I have read and understand the contents of this Statistical Analysis Plan, Version 2.0 for Study G1T28-212 dated 18 April 2023 and I agree with all the statistical approaches, variable derivations and data presentation detailed as described in this document.



# TABLE OF CONTENTS

| STATIS | TICAL ANALYSIS PLAN | 1 |
|---|---|---|
| SAP SIG | GNATURE PAGE | 2 |
| LIST O | F ABBREVIATIONS | 6 |
| 1. | INTRODUCTION | 8 |
| 1.1. | Study Design | 8 |
| 1.2. | Study Objectives | 10 |
| 1.3. | Sample Size Consideration | 10 |
| 2. | THE NUMBER OF PLANNED ANALYSES | 12 |
| 3. | ANALYSIS POPULATIONS | 13 |
| 3.1. | The Full Analysis Set – 1 (FAS1) | 13 |
| 3.2. | The Full Analysis Set – 2 (FAS2) | 13 |
| 3.3. | The Full Analysis Set (FAS) | 13 |
| 4. | GENERAL CONSIDERATIONS FOR DATA SUMMARY AND DISPLAY | 14 |
| 4.1. | Treatment Group Descriptions and Display in Table, Listings and Figures | 14 |
| 4.2. | Data Summary and Precision. | 14 |
| 4.3. | Definitions for Analysis Related Timepoint and Time Interval | 14 |
| 4.4. | Study Day | 15 |
| 4.5. | General Principles of Missing Data Handling | 16 |
| 5. | DISPOSITION AND BASELINE CHARACTERISTICS | 17 |
| 5.1. | Patient Disposition | 17 |
| 5.2. | Demographics and Baseline Disease Characteristics | 18 |
| 5.3. | Medical/Surgical History and Ongoing Conditions | 18 |
| 5.4. | Prior and Concomitant Medications | 18 |
| 5.5. | Summary of Protocol Deviations | 20 |
| 5.5.1. | Definitions and Process for Identifying Protocol Deviations | 20 |
| 5.5.2. | Summary of Protocol Deviations | 20 |
| 6. | CLASSIFICATION OF PRIOR SURGERIES AND PROCEDURES | 21 |
| 7. | STUDY DRUG EXPOSURE, DOSE INTENSITY AND MODIFICATION | 22 |
| 7.1. | Duration of Study Drug Exposure | 22 |
| 7.2. | Cumulative Dose and Dose Intensity | 22 |

| 7.3. | Study Drug Modifications | 24 |
|---|---|---|
| 8. | EFFICACY ANALYSIS | 26 |
| 8.1. | Definitions of Efficacy Endpoints | 26 |
| 8.1.1. | Primary Efficacy Endpoints – Change in CD8+ TILs/Tregs ratio from baseline to 7 ± 1 days after single-dose monotherapy trilaciclib administration | |
| 8.1.2. | Secondary Efficacy Endpoints – Pathologic complete response (pCR) rate at the time of definitive surgery | 26 |
| 8.1.3. | Exploratory Endpoints | 27 |
| 9. | SAFETY ANALYSIS | 28 |
| 9.1. | General Consideration of Safety Analysis | 28 |
| 9.2. | Adverse Events | 28 |
| 9.2.1. | Definition and Classification of Adverse Events | 28 |
| 9.2.2. | Imputation Rules for Missing Start or Stop Date for Adverse Events | 29 |
| 9.2.3. | Analysis for Adverse Events | 30 |
| 9.3. | Clinical Laboratory Data | 31 |
| 9.3.1. | Laboratory Parameters | 31 |
| 9.3.2. | Analysis for Laboratory Parameters | 32 |
| 9.4. | Vital Signs | 33 |
| 9.4.1. | Vital Sign Parameters | 33 |
| 9.4.2. | Analysis for Vital Signs | 34 |
| 9.5. | ECOG Performance Status | 34 |
| 9.6. | 12-lead Electrocardiograms | 34 |
| 9.6.1. | Electrocardiograms Parameters | 34 |
| 10. | CHANGES FROM THE PROTOCOL | 35 |
| 11. | REFERENCES | 36 |
| 12. | APPENDICES | 37 |
| APPEND | IX 1. SCHEDULE OF ASSESSMENTS | 38 |
| APPEND | IX 2. CUSTOMIZED MEDDRA QUERIES FOR TRILACICLIB AESIS | 40 |
| APPEND | IX 3. ANALYTICAL PLAN FOR QUANTIFICATION OF CD8+ TIL AND FOXP3+ CFLLS | 46 |

| | LIST OF TABLES | |
|---|---|---|
| Table 1: | Primary and Secondary Objectives and Endpoints | 10 |
| Table 2: | Statistical Power Calculation of Primary Endpoint | 11 |
| Table 3: | Definitions for Timepoints, Timepoint Related Assessments and Time Intervals | 15 |
| Table 4: | Dose Administration Parameters for Study G1T28-212 | 23 |
| Table 5: | Protocol Permitted Dose Reduction by Study Drug | 24 |
| Table 6: | Hematologic Preferred Terms to be Collapsed | 28 |
| Table 7: | Laboratory Categories and Parameters | 31 |
| Table 8: | Criteria for Potentially Clinically Significant Vital Signs | 33 |
| | LIST OF FIGURES | |
| Figure 1: | G1T28-212 Study Design Diagram | 9 |

# LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|--------------|------------------------------------------------|
| AC | anthracycline/cyclophosphamide |
| AE | adverse event |
| AESI | adverse event of special interest |
| ALT | alanine aminotransaminase |
| AST | aspartate aminotransferase |
| AUC | area under the plasma concentration-time curve |
| CD8+ | cluster of differentiation 8 positive |
| CDK | cyclin-dependent kinase |
| CI | confidence interval |
| COVID-19 | coronavirus disease 19 |
| CTCAE | Common Terminology Criteria for Adverse Events |
| ECG | electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | electronic case report form |
| EOS | End of study |
| FAS | Full Analysis Set |
| FOXP3 | Forkhead Box P3 |
| ICF | informed consent form |
| IFN | interferon |
| IHC | immunohistochemistry |
| INR | international normalized ratio |
| IV | intravenous |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MOA | mechanism of action |
| mRNA | messenger ribonucleic acid |
| MUGA | multigated acquisition |
| NCI | National Cancer Institute |

| Abbreviation | Definition |
|--------------|-------------------------------------------|
| pCR | pathologic complete response |
| PCS | potentially clinically significant |
| PD-L1 | programmed death-ligand 1 |
| PR | progesterone receptor |
| PT | Preferred term |
| Q1 | 25 <sup>th</sup> percentile |
| Q3 | 75 <sup>th</sup> percentile |
| Q3W | every 3 weeks |
| RBC | red blood cell |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SFU | Safety Follow-up |
| SOC | System organ class |
| TEAE | treatment-emergent adverse event |
| TIL | tumor-infiltrating lymphocyte |
| TNBC | triple negative breast cancer |
| Tregs | regulatory T cell |
| ULN | upper limit of normal |
| WHO-DD | World Health Organization Drug Dictionary |

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) provides detailed statistical methods, variable definitions and derivations, and data handling that will be applied to analyze the clinical trial data collected during study G1T28-212, "A Phase 2, Open-Label, Single-Arm Study of Single-Dose Lead-In and Neoadjuvant Trilaciclib and Chemotherapy in Patients with Early-Stage Triple Negative Breast Cancer (TNBC)" based on the protocol Version 2.0.

The Statistical Programming Supportive Documents (SPSD) will be developed based on the SAP to serve as companion documents of the SAP to guide programming realization of the SAP. The SPSD contain three separate documents:

- 1. The table of contents (TOC) for planned analyses (in Excel Spreadsheet).
- 2. The reporting conventions (in Word).
- 3. The shells or specificities for tables, listings, and figures (TLFs) generation (in Word).

If there are differences between statistical analysis approaches described in this SAP and those in the protocol, the methods and approaches in this SAP will supersede those in the protocol.

Changes and additions to the last signed off version of this SAP will be documented with corresponding rationale in the clinical study report (CSR).

Statistical software SAS® (SAS Institute Inc., Cary, NC) Version 9.4 or later will be used to perform data analyses following the plan as laid out in this SAP.

#### 1.1. Study Design

This is a Phase 2 multicenter, open-label, single-arm, neoadjuvant study with 4 phases:

- 1. Screening Phase,
- 2. Trilaciclib Lead-in Phase,
- 3. Treatment Phase, and
- 4. Surgery and Safety Follow-Up Phase.

During the Screening Phase, tumor tissue (sample #1) will be obtained at baseline prior to any study drug. This sample may be archival tissue, or if unavailable/insufficient, then a fresh biopsy is required. Patients with adequate archival tissue will also have the option to undergo an additional fresh biopsy at baseline. Patients will receive a single dose of monotherapy trilaciclib 240 mg/m² in the Trilaciclib Lead-in Phase, followed by tumor biopsy (sample #2) 7 (±1) days later. Following the biopsy, patients will enter the Treatment Phase in which trilaciclib 240 mg/m² on Day 1 of each cycle will be administered along with dose-dense anthracycline/cyclophosphamide followed by weekly taxane chemotherapy (doxorubicin 60 mg/m² + cyclophosphamide 600 mg/m² [AC] every 2 weeks for 4 cycles [Cycles 1-4], then weekly paclitaxel [T] 80 mg/m² weekly for 12 cycles [Cycles 5-16]). If pembrolizumab is given (per Investigator discretion), it will start with AC (Cycle 1 of chemotherapy). If carboplatin is given (per Investigator discretion) it will start with paclitaxel (Cycle 5).

Three to 5 weeks after the last dose of chemotherapy, patients will proceed to definitive surgery at which time tumor tissue (sample #3) will be collected if the patient has residual disease. A 30-day Safety Follow-up Visit will occur 30 (+7) days after the last dose of trilaciclib and an End of

Study Visit will occur within 14 days after surgery. Both the Safety Follow-up Visit and End of Study Visit may be conducted in person or by telephone and may occur on the same visit.

Figure 1: G1T28-212 Study Design Diagram



AC=doxorubicin/cyclophosphamide; C=cycle; Cb=carboplatin; D=day; Mono=monotherapy; Pembro=pembrolizumab; Q3W=every 3 weeks; QW=every week; SOC=standard of care; T=paclitaxel; TNBC=triple-negative breast cancer; Trila=trilaciclib; Tx=treatment

## 1.2. Study Objectives

#### **Primary:**

To evaluate the immune-based mechanism of action of trilaciclib after a single-dose as measured by the change in cluster of differentiation 8 positive (CD8+) tumor-infiltrating lymphocytes (TILs)/regulatory T cell (Tregs) ratio in tumor tissue.

## **Secondary:**

- To assess the pathologic complete response (pCR) rate at the time of definitive surgery.
- To evaluate the safety and tolerability of trilaciclib in combination with standard neoadjuvant systemic therapies.

Specifically, the primary and secondary objectives and their associated endpoints are described in Table 1.

**Table 1: Primary and Secondary Objectives and Endpoints** 

| Objectives | Endpoints |
|---|---|
| Primary Objective | |
| To evaluate the immune-based mechanism of action of trilaciclib after a single-dose as measured by the change in CD8+ TILs/Tregs ratio in tumor tissue | Change in CD8+ TILs/Tregs ratio in tumor tissue<br>from baseline to 7 days after single-dose<br>monotherapy trilaciclib administration |
| Secondary Objectives | |
| To assess the pCR rate at the time of definitive surgery | Rate of pCR using the definition of ypT0/Tis ypN0 (i.e., no invasive residual tumor in breast or nodes; noninvasive breast residuals allowed) as assessed by the local pathologist |
| To evaluate the safety and tolerability of trilaciclib in combination with standard neoadjuvant systemic therapies | Safety/tolerability as per CTCAE version 5.0 |

CD8+=cluster of differentiation 8 positive; CTCAE=Common Terminology Criteria for Adverse Events; pCR=pathologic complete response; TIL=tumor-infiltrating lymphocyte; Tregs=regulatory T cells

Other objectives and endpoints of the study can be found in Section 5 of the study protocol.

#### 1.3. Sample Size Consideration

Sample size justification is based off of previously published data on the CD8+/Tregs ratio from early stage TNBC patients who underwent neoadjuvant chemotherapy (Ahn). Using a 2-sided significance level of 0.05, and anticipating that 10% patients enrolled to this study will not have paired data (resulting in 27 patients with paired data), the power of the study to detect a

respective mean of paired difference in CD8+/Tregs ratio using paired Wilcoxon signed-rank tests has been calculated using PASS 2019 (v19.0.3), and is presented in Table 2.

**Table 2:** Statistical Power Calculation of Primary Endpoint

| Mean of Paired Difference in CD8+/Tregs | Power |
|---|---|
| 1.8 | 72% |
| 2.0 | 81% |
| 2.3 | 90% |
| 2.5 | 94% |
| Based on the assumption of an estimated standard deviation of paired differences of 3.4. | |

## 2. THE NUMBER OF PLANNED ANALYSES

There is only one planned analysis for this study. The planned analysis will be conducted to evaluate the immune-based mechanism of action of trilaciclib after a single dose as measured by the change in CD8+ TILs/Tregs ratio in tumor tissue. In addition, the pCR rate, at the time of definitive surgery as well as the safety and tolerability of trilaciclib in combination with standard neoadjuvant systemic therapies will be assessed.

#### 3. ANALYSIS POPULATIONS

# 3.1. The Full Analysis Set – 1 (FAS1)

The Full Analysis Set – 1 (FAS1) population includes enrolled patients who have received trilaciclib during the Trilaciclib Lead-in Phase. This population will be used to assess immune response in tumor tissue.

## 3.2. The Full Analysis Set -2 (FAS2)

The Full Analysis Set -2 (FAS2) population includes enrolled patients who have received at least one dose of any study drug during the Treatment Phase of the study.

#### 3.3. The Full Analysis Set (FAS)

The Full Analysis Set (FAS) population includes enrolled patients who received at least one dose of any study drug during the treatment period, where treatment period consists of the Trilaciclib Lead-in Phase and the Treatment Phase. This population will be used to assess safety and tolerability and the rate of pCR for trilaciclib in combination with neoadjuvant systemic therapies.

#### Version: 2.0

#### 4. GENERAL CONSIDERATIONS FOR DATA SUMMARY AND DISPLAY

# 4.1. Treatment Group Descriptions and Display in Table, Listings and Figures

This is a single-arm study in which all patients are treated with trilaciclib along with dose-dense anthracycline/cyclophosphamide followed by taxane chemotherapy (with optional administration of pembrolizumab and carboplatin). For TLFs that will be generated following SAP execution, the term *overall* will be used to describe all patients enrolled or all patients enrolled who have had at least one dose of any study drug, as applicable.

## 4.2. Data Summary and Precision

#### **General Principles of Data Summary**

Data will be summarized in table format for the respective analysis populations described in Analysis Populations. In general, continuous variables will be summarized based on number of patients with non-missing data (indicated by n), by mean, standard deviation (SD), median, Q1, Q3, minimum, and maximum values. Categorical variables will be summarized by number (n) and percentage of patients in each category.

# **General Principle of Data Listing**

All collected data and derived variables will be included in patient data listings. An indicator will be provided for any imputed data element (e.g., imputed adverse event [AE] onset date). Columns in listings will be ordered by study site, patient identification (ID), visit, and assessment or event date, if applicable, and then data elements.

#### General Principle of Precision for Summary Statistics and Calculated Statistical Quantities

The precision of summary statistics for continuous variables, including mean, median, Q1, Q3, minimum, and maximum, will be consistent with the precision of the variable as collected. Calculated quantities of variability (e.g., standard deviation, standard error [SE]) will be presented with one more decimal place than the precision of the variable that is collected. The boundaries of a confidence interval (CI) will keep the same precision as the point estimate.

When the collected data are integers (including counting variables), the mean, median, Q1, and Q3 will be presented with one decimal place.

For percentages, 1 digit will be presented after the decimal point (e.g., 10.1%). A percentage value less than 0.1% will be displayed as "<0.1%." A percentage value that is >99.9% and <100% will be displayed as ">99.9%."

P-values, in general, will be displayed in 3 decimal places except for when a p-value is less than < 0.001, it will be presented as "<0.001". If a p-value is greater than 0.999, it will be displayed as ">0.999".

Rounding will take place after all calculation steps are completed prior to result display.

## 4.3. Definitions for Analysis Related Timepoint and Time Interval

Timepoint and time intervals related to efficacy and safety data collected during the study will be summarized. For each specific category of data, the time interval by which the data will be

analyzed or summarized will be specified in the respective section in which the data analysis plan is described.

To clarify data inclusion for each time interval of interest and baseline or end values for each given time interval, Table 3 presents definitions for timepoints, timepoint related assessments, and time intervals involved in statistical data analysis or summary.

Table 3: Definitions for Timepoints, Timepoint Related Assessments and Time Intervals

| Term | Definition |
|---|---|
| Start of study (date) | Date of first dose of any study drug. |
| Study baseline | The last non-missing value prior to or on the date of the first dose of any study drug at the time that is before the time of the first study drug administration. If the event occurs on the same day as date of first dose of study drug but does not have the exact time captured, the event is assumed to have occurred prior to the first dose of study drug. |
| Pre-trilaciclib | The period before lead-in monotherapy trilaciclib administration when the first tumor biopsy (sample #1) will be obtained |
| Post-trilaciclib | The date that is $7 (\pm 1)$ days after lead-in monotherapy trilaciclib administration when the second tumor biopsy (sample #2) is obtained |
| Day 1 of Cycle X (date) | The date, during the Treatment Phase, when the first dose of any study drug for cycle X is administered. |
| End of cycle (date) | The date of Day 1 of the subsequent cycle, if there is a subsequent cycle. The end of the last cycle is the date of Safety Follow-up visit. If Safety Follow-up visit does not occur for a patient after the last dose of study drug, the End of cycle for the patient will be defined as 30 days post the last dose of study drug. |
| Duration of a cycle (days) | Total number of days from Day 1 of the cycle to End of cycle, that is, End of cycle – Day 1 of the cycle + 1. |
| Duration of study drug exposure (weeks) | The duration (in weeks) between the date of lead-in dose of monotherapy trilaciclib and End of the last cycle in the study. That is, (End of the last study cycle – Day 1 of lead-in dose of monotherapy trilaciclib + 1) / 7. |

# 4.4. Study Day

Study Day will be calculated for an event date or an assessment date to provide additional information for interpretation of the event occurrence. Study Day is calculated as:

• The start date of the event (visit date, onset date of an event, assessment date etc.) – date of first dose of any study drug + 1, if the event occurred on or after the reference date.

• The start date of the event (visit date, onset date of an event, assessment date etc.) – date of first dose of any study drug, if the event occurred prior to the reference date.

# 4.5. General Principles of Missing Data Handling

For primary efficacy endpoint the observed data are used for data summary and analyses. That is, no missing imputation will be performed. However, imputation of missing onset or stop dates for AEs and concomitant medication will be adapted to determine the status of each AE and the prior/concomitant/subsequent status of each non-study treatment medication. Please refer to 9.2.2 for the rules of imputation of missing AE onset or stop date and 5.4 for the rules of imputation of missing medication onset or stop dates.

For demographic and baseline characteristics, continuous variables will be summarized based on non-missing observations with the sample size of patients with non-missing data indicated, and a category of "Missing" will be included in the summary for each categorical variable.

#### 5. DISPOSITION AND BASELINE CHARACTERISTICS

### **5.1.** Patient Disposition

A summary of patient disposition will be generated using all accumulated data as of the database lock date.

In general, patient disposition summary will include the following 4 major sections:

- 1. Disposition of all screened patients who signed informed consent
- 2. Study drug disposition for patients who received at least one dose of any study drug
- 3. Study disposition for patients who were enrolled
- 4. Deaths among patients who were enrolled

The specific details for each section are described below.

# 1. Disposition of all screened patients

The total number of screened patients who signed informed consent will be presented as two mutually exclusive groups: those who were screen failures and those who were enrolled. For those who were enrolled, patients who received no study drug and those who receive a single dose of monotherapy trilaciclib during the Lead-in Phase are presented overall. Further, among patients who received a single dose of monotherapy trilaciclib, the number who had at least one dose of any study drug during the Treatment Phase will be summarized. Unless otherwise stated, number of enrolled patients will be the denominator for calculating percentages of patients in each of the categories.

#### 2. Study drug disposition

For each study drug (trilaciclib, doxorubicin, cyclophosphamide, pembrolizumab, paclitaxel and carboplatin), the number and percentage of patients who had at least one dose will be summarized. In addition, the number of patients who were discontinued from the study drug will be summarized. The number of patients who received at least one dose of study drug will be the denominator for the percentage calculation of number of patients who discontinued for the respective drug. For patients who discontinued the study drug, the primary reasons for study drug discontinuation will be presented with the percentage of patients in each reason being calculated based on the number of patients who discontinued the study drug.

#### 3. Study disposition

The number and percentage of patients who discontinued from the study will be summarized. The number of patients who were enrolled will be the denominator for the percentage calculation. The primary reason for study discontinuation will also be summarized, and the number of patients who discontinued the study will be the denominator for the percentage calculation for each reason of discontinuation.

#### 4. Death

The number and percentage of patients who died during the study will be summarized overall for all enrolled patients along with the primary reason of death (Progressive Disease, Adverse Event, Other). The number of enrolled patients will be the denominator for calculating percentages of

death, and the number of patients who died will be the denominator for calculating the percentage of patients within each reason for death.

Study drug and study disposition information will be provided in data listings for all enrolled patients.

#### 5.2. Demographics and Baseline Disease Characteristics

Demographics and baseline disease characteristics will be summarized on the FAS population.

Demographics including age at screening visit, age group (18-65, > 65), sex at birth, child-bearing potential, ethnicity, and race will be summarized. In addition, baseline body mass index (BMI) and Eastern Cooperative Oncology Group (ECOG) score will be summarized. Further, baseline disease characteristics such as stage at diagnosis, histologic grade, histopathological type at diagnosis, BRCA mutation and PD-L1 status will be summarized for all patients in the FAS population.

Data listing for demographics and baseline disease characteristics will be provided for all enrolled patients.

# 5.3. Medical/Surgical History and Ongoing Conditions

Surgical history and medical history and ongoing medical conditions at the Screening Visit will be summarized on the FAS population.

Non-breast cancer related medical history and ongoing medical conditions as collected at the Screening Visit will be coded using Medical Dictionary for Regulatory Activities (MedDRA) version 25.1 or later, and then summarized overall. Medical history and ongoing conditions will be presented by system organ class (SOC) and preferred term (PT), with both SOC and PT sorted in descending frequency based on the overall column. A patient will only be counted once within a particular SOC (or PT) even if the patient had multiple conditions/diseases in the same SOC (or PT).

A data listing for medical history and ongoing medical conditions collected at the Screening Visit will be provided for all enrolled patients. In addition, a data listing for prior surgeries/procedures will be generated for all patients in the FAS population.

## 5.4. Prior and Concomitant Medications

A summary of concomitant, non-cancer medications will be generated on the FAS population. Prior medications will be presented in a data listing. All prior medications will be collected from 21 days prior to signing the informed consent form (ICF).

Concomitant medications are those protocol-permitted medications that were given during the time interval from informed consent through the End of Study Visit. Vaccinations administered within 90 days prior to the first dose of study drug through the End of Study Visit will also be included as concomitant medications. Medications collected through electronic case report forms (eCRFs) will be coded to Anatomical Therapeutic Classification (ATC) and PT, where applicable, using the most recent World Health Organization Drug Dictionary (WHO-DD) version WHODrug-Global-B3 202209.

Concomitant medications will be summarized by ATC and PT and presented in a descending order of frequency for ATC and PT within an ATC based on the overall group. If a patient took multiple medications within the same ATC, the patient will only be counted once for that ATC. Similar logic applies to PT summaries. The number and percentage of patients receiving any concomitant medications will be summarized overall.

### Handling of Missing Start and/or End Date for Medications Entered into EDC

Medications with incomplete start and/or end dates will be imputed according to the specifications described below. Those with incomplete start and/or end dates will be assumed to be concomitant if it cannot be shown that the medication was taken outside of the treatment period.

#### For completely missing or partially missing start dates:

- If the start date has month and year but day is missing, the first dose date will be used if the month and year is the same as the first dose date, otherwise, the first day of the month will be used.
- If the start date has year, but day and month are missing, then the first dose date will be used if the year is the same as the first dose date, otherwise January 1<sup>st</sup> will be used.
- If the start date is completely missing, then it will be imputed as the first dose date of study drug.

After the imputation, the imputed start date will be compared with corresponding stop date, if available. If the imputed start date is later than the stop date, the start date will be imputed with the stop date instead.

For completely missing or partially missing stop dates for concomitant medications that are not ongoing at the time of study database lock:

- If the stop date has month and year but day is missing, the last day of the month will be used.
- If the stop date has year, but day and month are missing, December 31st will be used.
- If the stop date is completely missing, the last dose date will be used.

After the imputation, the imputed stop date will be compared against the death date for patients who died. If the date is later than the death date, the date of death will be used to impute the stop date instead.

Prior and concomitant medications will be listed with an indicator for prior or concomitant among all patients in the FAS population.

### 5.5. Summary of Protocol Deviations

### 5.5.1. Definitions and Process for Identifying Protocol Deviations

Protocol deviation refers to situations where a patient's eligibility for study entry or a specific data collection deviate from the entry criteria or study procedure as specified in the protocol. Protocol deviation cases at the patient level with specific data elements of concern need to be summarized and reported in the CSR. Protocol deviations will be categorized as major or minor. Major protocol deviations are those that could affect the integrity of the data or adversely affect patients' safety. Criteria that define major or minor protocol deviations will be specified, documented, and signed off prior to study database lock. Specifically, a protocol deviation specifications document that describes the criteria defining major and minor protocol deviations, the categories of major protocol deviations, and the list of patients who had at least one protocol deviation case with the classification of major or minor will be created and signed off prior to study database lock.

# 5.5.2. Summary of Protocol Deviations

A protocol deviation summary will be generated for the final analysis.

The number and percentage of patients in the FAS population with protocol deviations will be tabulated for each of the following categories.

- Patients with at least one protocol deviation (major or minor)
- Patients with at least one major protocol deviation
- Patients with at least one protocol deviation in each of the major deviation categories

Protocol deviations will be listed with details and flags for major or minor for all enrolled patients.

#### 6. CLASSIFICATION OF PRIOR SURGERIES AND PROCEDURES

Prior surgeries and procedures refer to those treatments that patients received prior to the Screening Visit. Summaries of prior surgeries and procedures will be based on the FAS population. The number and percentage of patients with any surgeries and procedures will be summarized. In addition, the number and percentage of patients with any surgeries and procedures related to the disease under study will be summarized.

A data listing for prior surgeries and procedures collected at the Screening Visit will be provided for all patients in the FAS population.

#### 7. STUDY DRUG EXPOSURE, DOSE INTENSITY AND MODIFICATION

Analyses described in this section will be based on the FAS population unless otherwise specified.

## 7.1. Duration of Study Drug Exposure

Duration of study drug exposure (weeks) is defined as the duration from date of lead-in dose of monotherapy trilaciclib to date of End of cycle for the last cycle. That is, duration of study drug exposure (weeks) = (Date of End of cycle for the last cycle – date of lead-in dose of monotherapy trilaciclib + 1)/7, where the definition for End of cycle for the last cycle is provided in 4.3.

For each study drug, the number of patients who received the study drug at each cycle (including the Lead-in Phase) will be summarized. In addition, the total number of cycles that a patient received will be summarized as a continuous variable, as well as a categorical variable. That is, descriptive summary statistics will be provided for the total number of cycles that patients received, and the number and percentage of patients who received exactly 0, 1, 2..., to the maximum number of cycles will be summarized.

Corresponding data listings will be provided.

#### 7.2. Cumulative Dose and Dose Intensity

The definitions for cumulative delivered dose, delivered dose intensity, relative cumulative dose, and relative dose intensity at the patient level, along with other parameters involved in the calculation of these variables are presented in Table 4. All collected dose information will be used in the calculation.

The calculated cumulative delivered dose, delivered dose intensity, relative cumulative dose, and relative dose intensity will be summarized as continuous variables for each study drug.

All variables described in Table 4 will be included in the data listing except for the study drug administration schedule.

 Table 4:
 Dose Administration Parameters for Study G1T28-212

| Parameter | Meaning | Trilaciclib | Doxorubicin | Cyclophosphamide | Paclitaxel | Pembrolizumab | Carboplatin |
|---|---|---|---|---|---|---|---|
| administration | Drug dose and<br>schedule per<br>protocol | 240 mg/m <sup>2</sup><br>administered as single-<br>dose monotherapy in<br>Trilaciclib Lead-in<br>Phase, then on Day 1<br>of each chemotherapy<br>cycle | 60 mg/m <sup>2</sup> once every<br>2 weeks for 4 cycles<br>(Cycles 1-4) | 600 mg/m <sup>2</sup> once every<br>2 weeks for 4 cycles<br>(Cycles 1-4) | 80 mg/m <sup>2</sup> once every<br>week for 12 cycles<br>(Cycles 5-16) | 400 mg once every 6<br>weeks starting on Day<br>1 of Cycle 1 and<br>continue through<br>Treatment Phase | AUC 1.5 every week<br>starting on Day 1 of<br>paclitaxel chemotherapy<br>(Cycles 5-16) |
| | administered for | Sum of doses over the duration of trilaciclib administration [mg/m <sup>2</sup> ] | Sum of doses over the duration of doxorubicin administration [mg/m²] | Sum of doses over the duration of cyclophosphamide administration [mg/m²] | Sum of doses over the duration of paclitaxel administration [mg/m <sup>2</sup> ] | | Sum of doses over the<br>duration of carboplatin<br>administration<br>[AUC] |
| • | Cumulative dose<br>administered per<br>week | Cumulative delivered<br>dose / EXP<br>[mg/m²/week] | Cumulative delivered<br>dose / EXP2<br>[mg/m²/week] | Cumulative delivered<br>dose / EXP2<br>[mg/m²/week] | Cumulative delivered<br>dose / EXP3<br>[mg/m²/week] | Cumulative delivered<br>dose / (EXP2 + EXP3)<br>[mg/week] | Cumulative delivered<br>dose / EXP3<br>[AUC/week] |
| cumulative dose<br>(%) | (Cumulative<br>delivered dose /<br>Cumulative<br>prescribed dose)<br>×100 | [Cumulative delivered dose / (240 × (1+CYC+CYC2))] ×100 | [Cumulative delivered<br>dose / (60 × CYC)]<br>×100 | [Cumulative delivered dose / (600 × CYC)] ×100 | × CYC2)] ×100 | {Cumulative<br>delivered dose / [400<br>× CEL((EXP2 +<br>EXP3) / 6)]} ×100 | [Cumulative<br>delivered dose / (1.5<br>× CYC2)] ×100 |
| | (Delivered dose<br>intensity /<br>prescribed dose<br>intensity) ×100 | {Delivered dose<br>intensity / [(240 × (1 +<br>CYC + CYC2)) / (1 +<br>2CYC + CYC2)]}<br>×100 | ×100 | [Delivered dose intensity / (600/2)] ×100 | (Delivered dose<br>intensity / 80) ×100 | [Delivered dose<br>intensity / (400/6)]<br>×100 | (Delivered dose intensity / 1.5) ×100 |

AUC = area under curve; IV = intravenous; CYC = number of cycles during cycles 1-4; CYC2 = number of cycles during cycles 5-16; EXP = duration of study drug exposure in weeks including lead-in; EXP2 = duration of study drug exposure in weeks during cycles 1-4; EXP3 = duration of study drug exposure in weeks during cycles 5-16; CEL = ceiling (smallest integer ≥ the resulting decimal number)

### 7.3. Study Drug Modifications

Overall study drug modifications will be summarized on the FAS population. There are three types of study drug modification: dose reduction, cycle delay or infusion interruption. Protocol permitted dose reductions for each study drug are summarized in Table 5.

Version: 2.0

**Table 5:** Protocol Permitted Dose Reduction by Study Drug

| Study Drug | Maximum Number of Dose Reductions Allowed |
|------------------|-------------------------------------------|
| Trilaciclib | 0 |
| Doxorubicin | 2 |
| Cyclophosphamide | 2 |
| Paclitaxel | 2 |
| Carboplatin | 2 |
| Pembrolizumab | 0 |

The overall number of patients with any study drug modification will be summarized based on the FAS. In addition, study drug modifications will be summarized in each of the following categories: chemotherapy dose reduction, treatment cycle delay, and infusion interruption. The number and percentage of patients who had any chemotherapy dose reduction, any cycle delay, or any infusion interruption will be summarized.

More detailed summaries as outlined below will be provided.

**Dose reduction for a specific chemotherapy**. Four chemotherapies (doxorubicin, cyclophosphamide, paclitaxel, and carboplatin) can have dose reduction per protocol (Table 5). The number and percentage of patients who had at least one dose reduction during the treatment period will be summarized overall. Dose reduction is counting for all the reductions across these four study drugs during the treatment period. In addition, the number and percentage of patients in the following mutually exclusive categories: no chance to have any dose reduction (Cycle 1 treatment only), 0, 1, 2, up to the maximum number of reductions for the drug will be summarized. The reasons for dose reduction as collected in the eCRF will also be summarized for each of these chemotherapies.

<u>Cycle delay</u>. Information regarding whether a cycle was delayed was collected in the eCRF for each cycle. The number of cycles that have been delayed will be summarized as a continuous variable. In addition, the number and percentage of patients in each of the following mutually exclusive categories will be summarized: no chance to have any cycle delay (Cycle 1 treatment only), 0, 1, 2, and 3 or more cycle delays.

The reasons for cycle delay collected in eCRF are as follows:

- Low Neutrophil Count
- Low Platelet Count
- BOTH Low Neutrophil Count AND Low Platelet Count
- Other Hematologic Toxicity
- Non-hematologic toxicity
- Other

CONFIDENTIAL

The number and percentage of patients in each of the categories will be calculated based on the number of patients in the FAS population.

Infusion interruption. Infusion interruption was captured in the eCRF for each respective study drug with the reasons. In addition to summarizing the number and percentage of patients who had at least one infusion interruption for any study treatment, the summary statistics for the total number of infusion interruptions and the number and percentage of patients in each of the following mutually exclusive categories will be summarized: 0, 1, 2, and 3 or more infusion interruptions. The number of interruptions is the sum of infusion interruptions for all study drugs for which the interruption occurred at least once during the infusion across all cycles in the Treatment Phase and Trilaciclib Lead-in Phase. Multiple interruptions for a drug during an infusion will only be counted once. The reasons for infusion interruption as collected in the eCRF will also be summarized.

Corresponding data listings will be provided.

#### 8. EFFICACY ANALYSIS

The parameters needed for the primary immune-response measure – the ratio of CD8+ TIL over Forkhead Box P3 (FOXP3)+ regulatory T cells (abbreviated as CD8+ TILs/Tregs) will be measured by our bio-marker vendor and a detailed analytical plan for the quantification of CD8+ TILs and FOXP3 is included in Appendix 3. Briefly, CD8+ TILs and FOXP3+ cells will be quantitated on baseline and Day 7 tumor samples using two independent immunohistochemistry (IHC) assays, PanCK/CD8 IHC and FOXP3 IHC, respectively. The IHC slides are evaluated by a pathologist and the derived density (/mm2) of CD8+ TILs and FOXP3+ cells will be used to determine the ratio of CD8+ TILs/Tregs.

Version: 2.0

## 8.1. Definitions of Efficacy Endpoints

# 8.1.1. Primary Efficacy Endpoints – Change in CD8+ TILs/Tregs ratio from baseline to $7 \pm 1$ days after single-dose monotherapy trilaciclib administration

From biopsy samples (archival or fresh) obtained, the ratio of CD8+ TILs to Tregs will be calculated at pre-trilaciclib and post-trilaciclib. Among patient with paired results, the difference in the ratio from pre-trilaciclib to post-trilaciclib will be calculated as

$$\text{Change in } \left( \frac{\text{CD8 + TILs}}{\text{Tregs}} \right) = \left( \frac{\text{CD8 + TILs}}{\text{Tregs}} \right)_{post-trilaciclib} - \left( \frac{\text{CD8 + TILs}}{\text{Tregs}} \right)_{pre-trilaciclib}$$

For patients with missing value at baseline or day 7, no imputation will be carried out.

Histograms and Box plot for the distribution of the change in CD8+ TILs/Tregs will be generated. In addition, a scatter plot for the correlation between pre and post trilaciclib ratio of CD8+ TILs/Tregs will also be generated.

The change in the ratio of CD8+ TILs to Tregs will be categorized as positive (change in [CD8+ TILs/Tregs] > 0), negative (change in [CD8+ TILs/Tregs] < 0), unchanged (change in [CD8+ TILs/Tregs] = 0) or not evaluable. Further, categories for the incremental units of 1.5 will be created for positive and negative changes. In situations where 2 or more consecutive units of 1.5 yield zero counts, such categories will be combined until the next unit of 1.5 with > 0 count.

Summary statistics for CD8+ TILs/Tregs among patients with both pre- and post-trilaciclib data will be provided for measurements taken at baseline (pre-trilaciclib),  $7 \pm 1$  days after single dose trilaciclib (post-trilaciclib), and the change scores (post minus pre). The significance of the magnitude of change will be compared using paired Wilcoxon Signed-Rank test. As sensitivity analysis, patients with neuroendocrine features of the disease will be excluded and the comparison analysis will be repeated.

The primary efficacy endpoint defined in this section will be derived based on FAS1 population.

# 8.1.2. Secondary Efficacy Endpoints – Pathologic complete response (pCR) rate at the time of definitive surgery

pCR will be evaluated using the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; residual noninvasive in breast allowed) as assessed by the local pathologist at the time

Version: 2.0

of definitive surgery. The pCR rate will be reported with a 95% confidence interval using the Clopper-Pearson method based on FAS population.

In addition, subgroup analyses will be conducted on the pCR rate by classifying patients into 2 distinct groups using the following criteria:

- High change in CD8+ TILs/Tregs from pre- to post-trilaciclib (> median value) vs. Low change in CD8+ TILs/Tregs from pre- to post-trilaciclib (\le median value).
- Positive vs. negative changes in CD8+ TILs/Tregs (unchanged CD8+ TILs/Tregs will be grouped with positive changes).

pCR rate will be summarized by subgroup and Fisher's exact test will be used to assess the association between pCR status and subcategories above.

Further, summary statistics for the change in CD8+ TILs/Tregs (from pre- to post-trilaciclib) will be provided for patients who had pCR and those who did not have pCR (pCR=Yes vs. pCR=No vs. pCR=Missing). Finally, where applicable, boxplots for the distribution of change in CD8+ TILs/ Tregs by pCR subcategories (Yes vs. No vs. Missing) will be presented.

The secondary efficacy endpoint defined in this section will be derived based on the FAS population.

#### 8.1.3. Exploratory Endpoints

The following endpoints will be explored. The description of the detailed steps involved in the analyses of these endpoints is outside the scope of this SAP.

- Immune-specific RNA profiling of tumor tissue at baseline, 7 days after single-dose monotherapy trilaciclib administration, and at surgery as quantified by CD8+ T cell and Tregs infiltration
- Longitudinal immune changes in peripheral blood, measured by frequency of immune subsets and profiling of activation, maturation, and exhaustion status
- Ex-vivo measurement of cytokine production to determine T cell function and polyfunctionality
- pCR in patients by subgroups (e.g., CDK4/6 dependence signatures: CDK4/6 dependent, CDK4/6 independent, CDK4/6 indeterminate; PD-L1 status as measured by IHC: positive, negative)
- pCR in patients by gene signatures identified in the tumor at baseline
- pCR in patients by frequency of immune subsets, immunological markers, and cytokines

#### 9. SAFETY ANALYSIS

## 9.1. General Consideration of Safety Analysis

Unless otherwise specified, all safety data collected during the study will be summarized. Hence, safety data summaries will be based on the FAS as defined in 3.3 of this SAP.

Version: 2.0

Safety data will be summarized using descriptive statistics for all patients when appropriate. All safety data collected through scheduled or non-scheduled visits during the study will be included in the safety data analyses. Missing safety data will generally not be imputed, unless otherwise specified.

Baseline assessment is, in general, defined as the last non-missing observation prior to receiving the first dose of any study drug.

#### 9.2. Adverse Events

#### 9.2.1. Definition and Classification of Adverse Events

AEs are defined as those AEs occurring on or worsening in severity after the first dose of any study drug (i.e., the conventional treatment-emergent AEs). Only AEs as described above are collected in the study database. All AEs are reported from the first dose of any study drug until end of study (EOS) visit. If EOS visit does not exist, then AEs until safety follow-up (SFU) visit date will be reported, if SFU date does not exist then AEs collected until, and including, 30 days after the last dose of study drug will be reported. SAEs thought to be related to a study specific procedure are also collected between the time the patient signs the informed consent and the first dose of any study drug.

AEs will be coded from verbatim text to PT and grouped by primary SOC according to MedDRA version 25.1. The severity (toxicity grades 1-5) of AEs will be graded according to the NCI CTCAE version 5.0 by the Investigator.

#### **Hematologic Adverse Events**

AEs related to hematologic toxicity will be collapsed based on the PTs from MedDRA version 25.1 and will be summarized separately (see 9.2.3). Table 6 outlines those PTs that will be collapsed.

Table 6: Hematologic Preferred Terms to be Collapsed

| Term presented in the Output | Preferred Term |
|------------------------------|--------------------------------|
| Neutropenia | Neutropenia |
| | Neutrophil count decreased |
| Anemia | Anemia |
| | Anaemia |
| | Red blood cell count decreased |
| | Hemoglobin decreased |

| Thrombocytopenia | Thrombocytopenia | Thrombocytopenia |
|------------------|----------------------------------|------------------|
| | Platelet count decreased | |
| Lymphocytopenia | Lymphocytopenia | |
| | Lymphopenia | |
| | Lymphocyte count decreased | |
| Leukopenia | Leukopenia | |
| | White blood cell count decreased | |

Version: 2.0

#### **Trilaciclib Adverse Events of Special Interest**

AEs of special interest (AESI) for trilaciclib have been identified, reflecting either the findings in the AEs from the previous studies of trilaciclib or class effects for CDK 4/6 inhibitors. AESI for trilaciclib will be identified by searching MedDRA PTs based on the Customized MedDRA Queries as detailed in Appendix 2.

Specifically, trilaciclib AESI include the following 5 categories:

- Injection site reaction/Phlebitis/Thrombophlebitis
- Acute drug hypersensitivity reaction
- Hepatotoxicity
- Interstitial lung disease /Pneumonitis
- Embolic and thrombotic events, venous

#### 9.2.2. Imputation Rules for Missing Start or Stop Date for Adverse Events

AEs with start/stop dates that are partially or completely missing that are not ongoing at the time of data cutoff will be imputed according to the specifications below in order to classify AEs.

For completely missing or partially missing AE start date:

- If the start date has month and year but day is missing, the first dose date will be used if the month and year is the same as the first dose date, otherwise, the first day of the month will be used.
- If the start date has year, but day and month are missing, then the first dose date will be used if the year is the same as the first dose date, otherwise January 1<sup>st</sup> will be used.
- If the start date is completely missing, then it will be imputed as the first dose date of study drug.

After the imputation, the imputed start date will be compared with AE stop date, if available. If the imputed start date is later than the stop date, the start date will be imputed with the stop date instead.

For completely missing or partially missing AE stop dates:

- If the stop date has month and year but day is missing, the last day of the month will be used.
- If the stop date has year, but day and month are missing, December 31st will be used.
- If the stop date is completely missing, then the date of EOS visit will be used; if EOS visit does not exist, then the SFU visit date is used, if SFU date does not exist then the last dose date + 30 days will be used.

After the imputation, the imputed AE stop date will be compared against the death date for patients who died. If the date is later than the death date, the date of death will be used to impute the stop date instead.

Every attempt will be made to obtain complete information for AEs regarding severity (i.e., CTCAE Grade) and relationship to drug. However, in the rare case of missing data, the following conservative approach will be taken for summary purpose. The non-imputed raw data will be presented in AE listings.

- Missing AE grade will be classified as 'Grade 3'
- Missing AE relationship will be classified as "Related"

### 9.2.3. Analysis for Adverse Events

AEs will be summarized by number and percentage of patients having at least one occurrence at the PT and SOC level overall. Patients with more than one occurrence of the same SOC (PT) will be counted only once within the SOC (PT) categorization. In general, the percentage of patients with an event will be calculated using the number of patients in the FAS as the denominator. For tables summarizing AEs related to study drugs the percentages will instead be calculated using the number of patients who received the drug as the denominator.

AEs will also be summarized by CTCAE grade and relationship to study drug (to any study drugs and to each individual study drug). Should a patient experience more than one occurrence of the same SOC (PT), the patient's worst occurrence (highest grade or highest related causality) will be used for the analysis and reporting.

In AE summaries, the SOC and PT within a SOC will be presented in descending order based on the incidence from all patients. If the incidence for two or more PTs is equal, these PTs will be presented in alphabetical order.

The AEs by decreasing frequency in PT during the trilaciclib Lead-in Phase will be summarized based on FAS1.

An overall AE summary table will be generated to present general information related to AEs including the following categories: number and percentage of patients with any AE, Serious AEs, AEs with CTCAE Grade  $\geq 3$  or 4, AEs leading to discontinuation of any study drug, AEs leading to death, AEs related to study drug (to any study drug, to trilaciclib, and to each other study drug).

In addition, the following summary tables will be generated, and they will be, in general, presented by SOC and PT unless otherwise specified.

- 1. AEs by decreasing frequency of PT during trilaciclib Lead-in Phase
- 2. AEs by decreasing frequency of PT during treatment period
- 3. AEs by PT and CTCAE Grade
- 4. AEs with CTCAE Grade 3 or 4 by PT
- 5. AEs leading to discontinuation of any study drug
- 6. AEs leading to death
- 7. AEs related to any and each study drug
- 8. Hematological AEs by collapsed PT and CTCAE grade
- 9. Serious AEs
- 10. Serious AEs related to any and each study drug
- 11. AESI for trilaciclib will be summarized.

In the above, hematological AEs will be reported using their coded PT with the exception of item 8 (Hematological AEs by collapsed PT and CTCAE grade), for which the collapsed terms as specified in Table 6 (9.2.1) will be reported in place of coded PT.

Corresponding AE listings will be provided to clearly indicate, at the patient level, the AE and SAE occurrence, start/stop date, relative study days to onset or stop, grade and causality for each AE. AESI for trilaciclib will also be listed with a similar level of detail. The AE listings will be generated based on FAS.

## 9.3. Clinical Laboratory Data

#### 9.3.1. Laboratory Parameters

Blood and urine samples for the determination of clinical chemistry, hematology, urinalysis and other laboratory variables described in Table 7 will be measured according to Schedule of Assessments in Appendix 1.

**Table 7:** Laboratory Categories and Parameters

| Lab Category | Lab Parameters |
|---|---|
| Hematology | white blood cell (WBC), platelets, hemoglobin, absolute neutrophil count (ANC). |
| Serum<br>Chemistry | Sodium, Potassium, Chloride, Bicarbonate, Urea, Phosphorus, Creatinine, Calcium, Magnesium, Total Protein, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Bilirubin, Albumin. |
| Coagulation | Prothrombin time and/or international normalized ratio |
| Urinalysis | Semiquantitative dipstick: specific gravity, pH, evaluation of glucose, protein, bilirubin, ketones, leukocytes, and hemoglobin |

| Microscopic examination (including RBC, WBC, and casts) will be performed if clinically warranted |
|---|
| Serum or urine human chorionic gonadotropin (hCG) pregnancy test (for WOCBP only) |

hCG=human chorionic gonadotropin; RBC=red blood cell; WBC=white blood cell; WOCBP=woman of childbearing potential

For hematology parameters, if absolute counts are not provided, those values will be derived from the differential percentage by multiplying differential percentage value with leukocyte value from the same sample. The normal ranges will be left missing in those cases.

Clinical chemistry and hematology assessments will be graded according to NCI CTCAE criteria, Version 5.0 or later. The determination of CTCAE grade for each measurement will be based on the collected laboratory values and will not involve clinical judgement. For laboratory parameters that CTCAE toxicity grade are not available, they will not be included in the analyses in which toxicity grades are reported. Instead, these parameter results will be classified and reported by the low/normal/high based on the laboratory normal reference ranges.

#### **Abnormal Hepatic Laboratory Values**

Abnormal hepatic laboratory values are defined in the following categories including any occurrence among all on-treatment, post-baseline assessments including scheduled and unscheduled values.

- Hy's Law: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 3x the upper limit of normal (ULN), alkaline phosphatase (ALP) < 2xULN, and total bilirubin  $\geq 2xULN$
- AST: > 3 and  $\le 5x$  ULN, > 5 and  $\le 8x$  ULN, > 8 and  $\le 10x$  ULN, > 10 and  $\le 20x$ ULN, and > 20x ULN; AST > 5x ULN for more than 5 weeks.
- ALT: >3 and  $\leq 5x$  ULN, > 5 and  $\leq 8x$  ULN, > 8 and  $\leq 10x$  ULN, > 10 and  $\leq 20x$ ULN, and > 20x ULN; ALT > 5x ULN for more than 5 weeks.
- Total bilirubin > 1.5xULN and < 2xULN,  $\ge 2$ xULN

#### 9.3.2. **Analysis for Laboratory Parameters**

Laboratory data from all central and local laboratories will be included in the analyses. Different laboratories are likely using slightly different normal reference ranges, which should not affect the planned analysis since they are all categorical and reported based on CTCAE toxicity grade or relationship to the normal ranges. The default convention for reporting of laboratory units will be standard international (SI) units. If a lab value is reported using an inequality symbol e.g., less than (<) a certain value, or greater than (>) a certain value, the given numeric value will be used in the summary. Data will be presented in listings with their inequality symbol.

For each parameter in the clinical chemistry and hematology laboratory group, respectively, CTCAE toxicity grading is used to classify patients into a toxicity grade from 1 to 4 for each timepoint assessment. The number and percentage of patients with highest grade will be

Version: 2.0

summarized for each grade from 1 to 4 and Grade 3-4, along with such summary for the value collected at baseline.

For the laboratory parameters that cannot be classified by CTCAE grade, the number and percentage of patients in the categories of treatment-emergent low or treatment-emergent high based on the normal reference range associated with the parameter will be summarized.

In addition, shift in CTCAE grade from baseline to the worst post-baseline value will be produced. The shift tables will include patients who had non-missing baseline and at least one non-missing post-baseline value for the parameter of interest.

The number and percentage of patients in each category of abnormal hepatic laboratory values will be summarized.

Laboratory parameters will be listed by the group of chemistry, hematology, coagulation, and other tests. In the data listing, flags that indicate the corresponding CTCAE grades and the classifications relative to the laboratory reference ranges will be included. In addition, a separate listing will be prepared for patients who met Hy's law.

#### 9.4. Vital Signs

## 9.4.1. Vital Sign Parameters

Vital signs including pulse rate, systolic blood pressure (SBP), diastolic blood pressure (DBP), weight and height will be measured according to Schedule of Assessments in Appendix 1.

Baseline vital signs refer to the measurements taken on the date of the first dose of any study drug (only if time of vital measurement is prior to the time of dosing) or, in the event vitals are not taken on the date of first dose of study drug, at the Screening visit. Post-baseline assessments refer to the measurements taken after the first dose of any study drug during the study. Change from baseline to the highest/lowest value across all post-baseline measurements for each vital sign parameter will be calculated. Patients who had a non-missing baseline and at least one non-missing measurement post-first dose for a given parameter will be included in the calculation.

Patients are classified with respect to the criteria of potentially clinically significant (PCS) findings of vital signs, which are defined by the highest/lowest value among post-baseline assessments and/or the change from baseline to the highest/lowest observed value. Details of PCS criteria for vital signs can be found in Table 8.

**Table 8:** Criteria for Potentially Clinically Significant Vital Signs

| Parameter | Direction | Highest/Lowest<br>Observed Value | Change from Baseline to the<br>Highest/Lowest Observed Value |
|---|---|---|---|
| SBP | High | ≥180 mmHg | Increase ≥40 mmHg |
| | Low | ≤90 mmHg | Decrease ≥40 mmHg |
| DBP | High | ≥105 mmHg | Increase ≥ 20 mmHg |
| | Low | ≤ 50 mmHg | Decrease ≥20 mmHg |
| Heart Rate | High | ≥ 120 bpm | Increase ≥40 bpm |

| | Low | ≤ 50 bpm | Decrease ≥40 bpm |
|--------|------|----------|------------------|
| Weight | High | | Increase ≥10% |
| | Low | | Decrease ≥10% |

bpm=beats per minute; DBP-diastolic blood pressure; SBP=systolic blood pressure

#### 9.4.2. Analysis for Vital Signs

Number and percentage of patients who meet any PCS criteria for each vital sign parameter as well as for each criterion will be summarized.

All observed vital sign values, change from baseline at each post-first dose assessment, and PCS flag will be listed.

#### 9.5. ECOG Performance Status

ECOG performance status was assessed at the Screening Visit and at Day 1 of each treatment cycle during the study.

A shift table that tabulates ECOG status at baseline and the worst status post first dose of any study drug will be generated.

All ECOG data will be included in data listing.

#### 9.6. 12-lead Electrocardiograms

# 9.6.1. Electrocardiograms Parameters

The standard 12-lead Electrocardiogram (ECG) will collect heart rate, PR interval, QRS interval, RR interval, and QT interval at screening visit only. Additional ECGs may be performed as clinically indicated at any time during the study (Appendix 1).

Since either QTcF or QTcB could be collected by different study sites, QTcF (using Fridericia's method) will be calculated from the QT and RR (converted from collected ms to sec) intervals based on the formula:

QTcF = Uncorrected QT/ (RR Interval)^1/3, if QT and/or RR are missing, the QTcF will be left as missing.

A summary table of ECG parameters at baseline will be generated. In addition, ECG data will be included in data listing.

## 10. CHANGES FROM THE PROTOCOL

In section 12.2 of the protocol, FAS1 and FAS2 are defined as the study populations. In this SAP, a FAS population is defined to ensure that safety data for patients who dropped from the study after receiving a single dose of trilaciclib in the Lead-in Phase are adequately captured and summarized where necessary. The FAS population also includes patients who did not receive the single dose of trilaciclib in the Lead-in Phase before proceeding to the Treatment Phase.

# 11. REFERENCES

Soomin Ahn, Yul Ri Chung, An Na Seo, Milim Kim, Ji Won Woo, So Yeon Park. Changes and prognostic values of tumor-infiltrating lymphocyte subsets after primary systemic therapy in breast cancer. PLoS One. 2020;15(5):e0233037.
## 12. APPENDICES

## APPENDIX 1. SCHEDULE OF ASSESSMENTS

| | Screening | | nciclib<br>n Phase | Treatment Phase | | | | | Definitive<br>Surgery | Safety<br>Follow-u<br>p Visit | End of<br>Study<br>Visit | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Single | | +/ | Doxoru<br>yclophos<br>- pembr<br><i>ech cycle</i> | sphami<br>olizum: | ab | Paclitaxel<br>+/- carboplatin b<br>+/- pembrolizumab b<br>Each cycle = 1 week | | | | |
| Protocol Activity | | dose<br>mono.<br>trila. | On-tx<br>biopsy | C1<br>D1 <sup>a</sup> | C2<br>D1 | C3<br>D1 | C4<br>D1 | C5 through C16<br>D1 | | | | |
| Visit Window | Up to 21 days prior to first dose | N/A | 7d ±1d<br>after<br>trila | N/A | ±2d | ±2d | ±2d | ±1d | 3-5 weeks following tx. | 30d (+7)<br>after last<br>trila dose | Within<br>14d<br>after<br>surgery | See Protocol<br>Section for<br>Additional<br>Details |
| Informed consent | X | | | | | | | | | | | Section |
| ER-/PR-/HER2- status | X | | | | | | | | | | | Section |
| Inclusion/ exclusion criteria | X | | | | | | | | | | | Section |
| Baseline characteristics and demographics | X | | | | | | | | | | | Section |
| Medical and surgical history | X | | | | | | | | | | | Section |
| Concomitant medications and procedures | X | X | | X | X | X | X | X (C5, 8, 11, 16 only) | X | X | X | Section |
| Complete physical exam | X | | | | | | | | | | | Section |

| | Screening | | nciclib<br>n Phase | Treatment Phase | | | Definitive<br>Surgery | Safety<br>Follow-u<br>p Visit | End of<br>Study<br>Visit | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Single | | +/ | Doxoru<br>yclophos<br>- pembr<br><i>ch cycle</i> | phami<br>olizum: | ab | Paclitaxel<br>+/- carboplatin <sup>b</sup><br>+/- pembrolizumab <sup>b</sup><br>Each cycle = 1 week | | | | |
| Protocol Activity | | dose<br>mono.<br>trila. | On-tx<br>biopsy | C1<br>D1 <sup>a</sup> | C2<br>D1 | C3<br>D1 | C4<br>D1 | C5 through C16<br>D1 | | | | |
| Visit Window | Up to 21 days prior to first dose | N/A | 7d ±1d<br>after<br>trila | N/A | ±2d | ±2d | ±2d | ±1d | 3-5 weeks following tx. | 30d (+7)<br>after last<br>trila dose | Within<br>14d<br>after<br>surgery | See Protocol<br>Section for<br>Additional<br>Details |
| Directed physical exam | | X | | X | X | X | X | X (C5, 8, 11, 16 only) | | | | Section |
| Vitals | X | X | | X | X | X | X | X | | | | Section |
| ECOG performance status | X | X | | X | | | | X (C5 and 16 only) | | | X | Section |
| Adverse event reporting | X | X | | X | X | X | X | X | X | X | X | Section |
| Hematology | X | X | | X | X | X | X | X | | | | Section |
| Serum chemistry | Х | X | | X | X | X | X | X | | | | Section |
| Coagulation (PT or INR) | X | | | | | | | | | | | Section |
| 12-lead ECG | X | | | | | | | | | | | Section Error! Reference |

| | Screening | | aciclib<br>n Phase | Treatment Phase | | | Definitive<br>Surgery | Safety<br>Follow-u<br>p Visit | End of<br>Study<br>Visit | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Single | | +/ | Doxoru<br>yclophos<br>- pembr<br><i>ch cycle</i> | sphami<br>olizum: | ab | Paclitaxel<br>+/- carboplatin b<br>+/- pembrolizumab b<br>Each cycle = 1 week | | • | | |
| Protocol Activity | | dose<br>mono.<br>trila. | On-tx<br>biopsy | C1<br>D1 <sup>a</sup> | C2<br>D1 | C3<br>D1 | C4<br>D1 | C5 through C16<br>D1 | | | | |
| Visit Window | Up to 21 days prior to first dose | N/A | 7d ±1d<br>after<br>trila | N/A | ±2d | ±2d | ±2d | ±1d | 3-5 weeks following tx. | 30d (+7)<br>after last<br>trila dose | Within<br>14d<br>after<br>surgery | See Protocol<br>Section for<br>Additional<br>Details |
| | | | | | | | | | | | | source not found. |
| Echocardiogram or<br>MUGA for LVEF<br>assessment | X | | | | | | | | | | | Section |
| Urinalysis | X | | | | | | | | | | | Section |
| Urine/serum HCG<br>(WOCBP only) | X | | | X | | | | X (C5, 11, 16 only) | | | | Section |
| | | | | Bio | marker | and Ef | ficacy A | Assessments | | | | |
| Blood samples for biomarkers | | X<br>(pre-<br>dose) | X (pre-<br>biopsy) | | X<br>(pre-<br>dose) | | | | X (-3 day) | | | Section |
| Tumor sample #1 (Baseline) | X | | | | | | | | | | | Section |
| Tumor sample #2 (On treatment) | | | X | | | | | | | | | Section |
| Tumor sample #3<br>(Surgery) | | | | | | | | | X | | | Section Error! Reference |

| | Screening | | aciclib<br>n Phase | Treatment Phase | | | | | Definitive<br>Surgery | Safety<br>Follow-u<br>p Visit | End of<br>Study<br>Visit | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Single | | +/ | Doxoru<br>yclophos<br>- pembr<br><i>ch cycle</i> | sphami<br>olizum: | ab | Paclitaxel<br>+/- carboplatin b<br>+/- pembrolizumab b<br>Each cycle = 1 week | | | | |
| Protocol Activity | | dose<br>mono.<br>trila. | On-tx<br>biopsy | C1<br>D1 <sup>a</sup> | C2<br>D1 | C3<br>D1 | C4<br>D1 | C5 through C16<br>D1 | | | | |
| Visit Window | Up to 21 days prior to first dose | N/A | 7d ±1d<br>after<br>trila | N/A | ±2d | ±2d | ±2d | ±1d | 3-5 weeks following tx. | 30d (+7)<br>after last<br>trila dose | Within<br>14d<br>after<br>surgery | See Protocol<br>Section for<br>Additional<br>Details |
| | | | | | | | | | | | | source not found. |
| pCR assessment | | | | | | | | | X | | | iouna. |
| per assessment | | L | | | L | Treat | tment | | 71 | | 1 | |
| | | X | | X | X | X | X | X | | | | Section Error! Reference source not |
| Trilaciclib | | | | | | | | | | | | found. |
| Doxorubicin/<br>cyclophosphamide | | | | X | X | X | X | | | | | Section Error! Reference source not found. |
| Paclitaxel | | | | | | | | X | | | | Section |
| Carboplatin AUC 1.5 (Investigator discretion) | | | | | | | | X | | | | Section |
| Pembrolizumab<br>(Investigator discretion) | | | | X | | | X | X (C9 and C15 only) | | | | Section Error! Reference source not found. |
| Definitive surgery | | | | | | | | | X | | | Section |

AUC=area under the curve; C=cycle; chemo=chemotherapy; d=day; ECG=electrocardiogram; ECOG=Eastern Cooperative Oncology Group; ER=estrogen receptor; HCG=human chorionic gonadotropin; HER2=human epidermal growth factor receptor 2; INR=international normalized ratio; LVEF=left ventricular ejection fraction; mono=monotherapy;

MUGA=multiple-gated acquisition; N/A=not applicable; pCR=pathologic complete response; PR=progesterone receptor; PT=prothrombin time; q2w=every 2 weeks; trila=trilaciclib; tx=treatment; WOCBP=women of childbearing potential

<sup>&</sup>lt;sup>a</sup> C1D1 may be the same day as the on-treatment biopsy, as long as the biopsy is done prior to initiation of chemotherapy.

<sup>&</sup>lt;sup>b</sup> Per Investigator discretion.

| <b>AESI Categories</b> | Pro | eferred Terms |
|---|---|---|
| | Administration site phlebitis | Periphlebitis |
| l | Application site phlebitis | Phlebitis |
| | Catheter site phlebitis | Phlebitis deep |
| | Chemical phlebitis | Phlebitis infective |
| | Infusion site phlebitis | Septic phlebitis |
| | Infusion site thrombosis | Thrombophlebitis |
| | Injection site phlebitis | Thrombophlebitis septic |
| | Injection site thrombosis | Thrombophlebitis superficial |
| | | Vascular access site thrombosis |
| | Administration related reaction | Infusion site erythema |
| | Administration site dermatitis | Infusion site hypersensitivity |
| | Administration site | T.C |
| | hypersensitivity | Infusion site pain Infusion site rash |
| | Administration site pain Administration site rash | |
| | Administration site recall | Infusion site reaction |
| Injection Site | reaction | Infusion site recall reaction |
| Reaction/ | Administration site urticaria | Infusion site urticaria |
| Phlebitis/ | Administration site vasculitis | Infusion site vasculitis |
| Thrombophlebitis | Application site dermatitis | Injection related reaction |
| | Application site hypersensitivity | Injection site dermatitis |
| | Application site pain | Injection site erythema |
| | Application site rash | Injection site hypersensitivity |
| | Application site recall reaction | Injection site pain |
| | Application site urticaria | Injection site rash |
| | Application site vasculitis | Injection site reaction |
| | Catheter site dermatitis | Injection site recall reaction |
| | Catheter site hypersensitivity | Injection site urticaria |
| | Catheter site pain | Injection site vasculitis |
| | Catheter site rash | Installation site urticaria |
| | Catheter site urticaria | instillation site hypersensitivity |
| | Catheter site vasculitis | instillation site pain |
| | Immediate post-injection reaction | instillation site rash |
| | Infusion related reaction | Skin reaction |
| | Infusion site dermatitis | Vessel puncture site rash |
| | | Vessel puncture site vesicles |
| Acute drug | Allergic bronchitis | Laryngitis allergic |
| hypersensitivity | Allergic cough | Laryngospasm |
| reaction | Allergic eosinophilia | Laryngotracheal oedema |

| <b>AESI Categories</b> | Pr | eferred Terms |
|---|---|---|
| | Chronic hepatitis | Hepatocellular injury |
| | Coma hepatic | Hepatotoxicity |
| | Drug-Induced Liver Injury | Immune-mediated hepatitis |
| | Hepatic failure | Liver disorder |
| | Hepatic infiltration eosinophilia | Liver injury |
| | Hepatic necrosis | Mixed liver injury |
| | Hepatic steato-fibrosis | Non-alcoholic steatohepatitis |
| | Hepatic steatosis | Steatohepatitis |
| | Hepatitis | Subacute hepatic failure |
| | Acute interstitial pneumonitis | Idiopathic interstitial pneumonia |
| | Acute lung injury | Idiopathic pneumonia syndrome |
| | Acute respiratory distress | |
| | syndrome | Idiopathic pulmonary fibrosis |
| | Alveolar lung disease | Immune-mediated pneumonitis |
| | Alveolitis | Interstitial lung disease |
| Interstitial Lung | Alveolitis necrotizing | Necrotizing bronchiolitis |
| Disease (ILD) | Autoimmune lung disease | Obliterative bronchiolitis |
| /Pneumonitis | Diffuse alveolar damage | Pneumonitis |
| | Eosinophilic pneumonia | Pneumonitis chemical |
| | Eosinophilic pneumonia acute | Progressive massive fibrosis |
| | Eosinophilic pneumonia chronic | Pulmonary fibrosis |
| | Granulomatous pneumonitis | |
| | Hypersensitivity pneumonitis | Pulmonary toxicity |
| | | Restrictive pulmonary disease |
| | Axillary vein thrombosis | Pulmonary thrombosis |
| | Brachiocephalic vein occlusion | Pulmonary vein occlusion |
| | Brachiocephalic vein thrombosis | Pulmonary veno-occlusive disease |
| | Deep vein thrombosis | Pulmonary venous thrombosis |
| | Embolism venous | Subclavian vein occlusion |
| Embolic and | Iliac vein occlusion | Subclavian vein thrombosis |
| thrombotic | Obstructive shock | Superior vena cava occlusion |
| events, venous | Pelvic venous thrombosis | Thrombosis |
| | Peripheral vein occlusion | Vena cava embolism |
| | Peripheral vein thrombus | |
| | extension | Vena cava thrombosis |
| | Phlebectomy | Venous occlusion |
| | Pulmonary embolism | Venous thrombosis |
| | Pulmonary microemboli | Venous thrombosis limb |

Venous thrombosis limb

Pulmonary microemboli

| Assay<br>Name | Tissue Type<br>(skin/tumor/) | Test SOP | Analysis SOP | Analysis Form | Remarks |
|---|---|---|---|---|---|
| PD-L1<br>SP142 IHC | Tumor | TE-IHC-198 | TE-IQ-16 | FO-390 | |
| PanCK/CD<br>8 IHC | Tumor | TE-IHC-153 | TE-IQ-36<br>TE-IQ-40 | FO-525<br>FO-526 | |
| CD8/FoxP3<br>/GZMB | Tumor | TE-IHC-246 | TE-IQ-137 | FO-760 | |
| FoxP3 | Tumor | TE-IHC-324 | TE-IQ-62 | FO-729 | |

PD-L1 SP142 will be scored according to SP142 algorithm (TE-IQ-16). The fraction of viable tumor cells (%) that express PD-L1 (discernible membrane staining of any intensity) can be scored. Cytoplasmic staining is not included in the scoring. In addition, immune cells are scored as a relative area estimate, i.e. the percentage of the tumor area that is covered by PD-L1-positive immune cells.

The PanCK-CD8 IHC slides will be evaluated by a pathologist for CD8 using the density proportion score algorithm (TE-IQ-40). The output of this analysis is the relative surface area (%) of the tumor with a CD8-positive immune cell density that belongs to one of the 8 density bins, and for each of the 8 density bins (8 data fields per IHC slide). The density bins are linked to reference images that are used by the pathologist. The reference images are marker-specific (CD8). There are 4 density bins (0-3) for intrastromal CD8-positive immune cells and 4 density bins (0-3) for intra-epithelial CD8-positive immune cells. In addition, the immune phenotype will be scored as 'desert', 'inflamed', 'excluded' in the PanCK-CD8 IHC slides based on the raw density proportion scores.

For the automated quantitative analysis (TE-IQ-36), a central tumor region is delineated by a pathologist. If an interface is present with adjacent normal tissue, an a 1000-µm wide invasive margin will be drawn. Visiopharm software is used to generate an epithelial carcinoma mask denoting the tumor region. The relative surface area (%) as well as density (#/mm²) of CD8-positive TILs can then be measured in both stromal and epithelial (carcinoma cell nests) compartments . If possible, these analyses will be performed for both the invasive margin and in the center of tumor samples. A 'tumor-stroma ratio' between the PanCK-positive carcinoma and the PanCK-negative stromal areas will be calculated, and areas will be provided for each region of interest.

CD8/GZMB/FoxP3 IHC will be scored according to TE-IQ-137. An assay to measure relative marker area and densities of CD8, FOXP3 and GZMB in solid tumor samples, within two regions of interest (ROIs): Central Tumor (CnTumor) and Invasive Margin (IM). The tumor region is delineated by a pathologist on the image of a serial HE-stained slide. The tumor annotation is copied manually onto the CD8-GZMB-FOXP3 image. If an interface is present with adjacent normal tissue, a 1000-µm wide invasive margin will be drawn. Single CD8-positive, single GZMB-positive, single FOXP3-positive, double CD8-GZMB-positive and double CD8-FOXP3-positive cells are automatically detected in the annotated regions through image analysis. The relative surface area (%) and density (#/mm²) of these different cell types can then be quantified as well as the proportion in relation to the CD8 population.

FoxP3-stained slides will be analyzed by the TE-IQ-62 method. A central tumor region is delineated by a pathologist. If an interface is present with adjacent normal tissue, an a 1000-µm wide invasive margin will be drawn. The relative area and the density of FoxP3-positive cells in central tumor and, if present, the invasive margin are quantified.